CLINICAL TRIAL: NCT03989076
Title: Evaluating the Mechanism of Changes to Inferior Vena Cava Diameter Using Point of Care Ultrasound in Patients Undergoing Interscalene Brachial Plexus Block
Brief Title: Inferior Vena Cava (IVC) Diameters Before & After Interscalene Block
Status: Withdrawn | Type: Observational
Why Stopped: unable to enroll subjects
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rodney Gabriel, Principal Investigator, University of California, San Diego
Other Study IDs: UCSD 181482
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: IVC - Inferior Vena Cava Abnormality

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Interscalene Brachial Plexus Block — Analgesic nerve block as part of routine care with pre- and post-block ultrasonographic imaging of the diaphragm and inferior vena cava
  Other Names: Point of Care Ultrasound

SUMMARY:
The purpose of this study is to understand how changes to breathing patterns in the chest affect blood flow to the heart from the inferior vena cava in the abdomen. Ultrasound of the upper abdomen will be used to visualize changes in breathing patterns in the chest and blood flow in the abdomen.

DETAILED DESCRIPTION:
In recent practice, point-of-care ultrasound has been used to assess the size and respiratory variation of the inferior vena cava as a marker for volume status and fluid responsiveness. Little investigation has occurred regarding the mechanism of observed respiratory variation. Anesthetic plans for surgery (e.g. shoulder replacement) frequently employ interscalene injections to target and block the brachial plexus, which (on the same side) results in phrenic nerve palsy and paralysis of the diaphragm. The goal of this study is to examine the relationship between diaphragmatic function and variation in IVC diameter. Specifically, the investigators will evaluate and compare the size and variability of the inferior vena cava by point-of-care ultrasound before and after brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age > 18 years)
* Scheduled to receive an interscalene block

Exclusion Criteria:

* Any person with known, pre-existing phrenic nerve, diaphragmatic, or inferior vena cava anomaly.
* Patients who cannot be successfully imaged by ultrasound or who cannot participate in spirometry will additionally be excluded.
* Non-English speaking patients will be excluded as well as there is no research funding to translate consent forms. Given that there is no potential benefit to participation in the study, this does not exclude these individuals from any potentially beneficial therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult (age > 18 years) patients undergoing surgery of any type at UC San Diego Medical Center for whom the surgeon has requested an interscalene nerve block and for whom the block is clinically indicated as determined by the primary anesthesiologist.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Ipsilateral hemiparesis | Within 30 minutes post-block
  Detectable paralysis of the ipsilateral hemidiaphragm by point of care ultrasound
IVC Collapsibility Index Change | Within 30 minutes post-block
  Measured IVC diameter and collapsibility by point of care ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Medical Center, La Jolla, California, United States

REFERENCES:
- [Background] Nagdev AD, Merchant RC, Tirado-Gonzalez A, Sisson CA, Murphy MC. Emergency department bedside ultrasonographic measurement of the caval index for noninvasive determination of low central venous pressure. Ann Emerg Med. 2010 Mar;55(3):290-5. doi: 10.1016/j.annemergmed.2009.04.021. Epub 2009 Jun 25. PMID 19556029
- [Background] Feissel M, Michard F, Faller JP, Teboul JL. The respiratory variation in inferior vena cava diameter as a guide to fluid therapy. Intensive Care Med. 2004 Sep;30(9):1834-7. doi: 10.1007/s00134-004-2233-5. Epub 2004 Mar 25. PMID 15045170
- [Background] Magder S. Bench-to-bedside review: An approach to hemodynamic monitoring--Guyton at the bedside. Crit Care. 2012 Oct 29;16(5):236. doi: 10.1186/cc11395. PMID 23106914
- [Background] Kimura BJ, Dalugdugan R, Gilcrease GW 3rd, Phan JN, Showalter BK, Wolfson T. The effect of breathing manner on inferior vena caval diameter. Eur J Echocardiogr. 2011 Feb;12(2):120-3. doi: 10.1093/ejechocard/jeq157. Epub 2010 Oct 27. PMID 20980326
- [Background] Gignon L, Roger C, Bastide S, Alonso S, Zieleskiewicz L, Quintard H, Zoric L, Bobbia X, Raux M, Leone M, Lefrant JY, Muller L. Influence of Diaphragmatic Motion on Inferior Vena Cava Diameter Respiratory Variations in Healthy Volunteers. Anesthesiology. 2016 Jun;124(6):1338-46. doi: 10.1097/ALN.0000000000001096. PMID 27003619
- [Background] El-Boghdadly K, Chin KJ, Chan VWS. Phrenic Nerve Palsy and Regional Anesthesia for Shoulder Surgery: Anatomical, Physiologic, and Clinical Considerations. Anesthesiology. 2017 Jul;127(1):173-191. doi: 10.1097/ALN.0000000000001668. PMID 28514241
- [Background] Boon AJ, Sekiguchi H, Harper CJ, Strommen JA, Ghahfarokhi LS, Watson JC, Sorenson EJ. Sensitivity and specificity of diagnostic ultrasound in the diagnosis of phrenic neuropathy. Neurology. 2014 Sep 30;83(14):1264-70. doi: 10.1212/WNL.0000000000000841. Epub 2014 Aug 27. PMID 25165390